CLINICAL TRIAL: NCT03071926
Title: Efficacy and Safety of Metronomic Pegylated Liposomal Doxorubicin in Patients With Primary Endocrine Resistant Advanced Breast Cancer
Brief Title: Metronomic PLD in Patients With Primary Endocrine Resistant ABC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Vice Director of department of medical oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2017-22
Record Dates: First submitted 2017-02-27; First posted 2017-03-07 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pegylated Liposomal Doxorubicin (Experimental): Pegylated Liposomal Doxorubicin: 20 mg, qw, first 6 weeks ,every 8 weeks
  Interventions: Drug: Pegylated Liposomal Doxorubicin

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin — 20 mg, qw, first 6 weeks ,every 8 weeks

SUMMARY:
Metronomic PLD in Patients with Primary Endocrine Resistant ABC

DETAILED DESCRIPTION:
Efficacy and Safety of Metronomic Pegylated Liposomal Doxorubicin in Patients with Primary Endocrine Resistant Advanced Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 and 75 years old
2. ECOG: 0～2
3. Life expectancy longer than 3 months
4. Histological proven unresectable recurrent or metastatic HR positive/HER2 negative breast cancer
5. Primary endocrine resistance is defined as: a relapse while on the first 2 years of adjuvant ET, or PD within first 6 months of first-line ET for MBC, while on ET
6. At least one measurable disease according to RECIST 1.1(except for bone metastasis only)
7. LVEF ≥ 55%
8. No radiation therapy within 4 weeks prior to enrollment
9. Normal function of major organs: Hb ≥ 90 g/L (no blood transfusion within 14 days) ;ANC ≥1.5×109 /L；PLT ≥75×109 /L；TBIL≤1. 5×ULN; ALT、 AST≤ 3×ULN（ALT、 AST≤ 5×ULN with hepatic metastases）; serum Cr ≤ 1×ULN
10. Be willing to participate in the study, sign informed consent and cooperate with the follow-up

Exclusion Criteria:

1. Previous accumulated or equivalent dose of doxorubicin ≥300mg/m2
2. Intervals of anthracycline-based adjuvant chemotherapy ≤1 year (time between anthracycline-based adjuvant or neoadjuvant chemotherapy and disease relapse)
3. Patients with symptomatic central nervous system metastases. Except for patients with stable and asymptomatic brain metastases for at least 8 weeks and no need for glucocorticoids or mannitol treatment before the trial and at least one measurable lesion outside the brain. Radiotherapy for brain metastases should be completed at least 4 weeks before the registration
4. Pregnant or lactating women and gestational age women who are unable to use effective contraception
5. Treatment with investigational products within 4 weeks before the study
6. Severe cardiopulmonary insufficiency, severe hepatic and renal dysfunction
7. Severe or uncontrolled infection
8. Psychiatric drugs abuse and unable to withdrawal or mental disorders
9. Other malignancies, except for cured skin basal cell carcinoma and cervical intraepithelial neoplasia.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression Free Survival

SECONDARY OUTCOMES:
Number and grade of treatment-related cardiotoxicity as assessed by CTCAE v4.0 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  monitoring LVEF
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall Survival
CBR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Clinical Benefit Rate

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China